CLINICAL TRIAL: NCT02460406
Title: The Effects of Lower Limb Progressive Functional Strength Training Protocol on Body Functions and Activity in Children With Unilateral Spastic Cerebral Palsy: a Single-blind Randomized Controlled Trial
Brief Title: Progressive Functional Strength Training in Unilateral Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, PT, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/224
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: strength training; virtual reality; plyometric exercises; cerebral palsy; hemiplegic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): traditional physiotherapy (stretching, normal range of movement, walking)
  Interventions: Other: traditional physiotherapy
- intervention group (Active Comparator): progressive functional strength training protocol on lower extremities consisted of functional squat system with virtual reality in leg press, plyometric exercises, exercises with Bosu ball & heel-rise exercises.
  Interventions: Other: progressive functional strength training

INTERVENTIONS:
Other: traditional physiotherapy — We are applying routine traditional physiotherapy consisted of neurodevelopmental treatment (stretching, weight bearing, functional reaching & walking so on).
  Arms: control group
Other: progressive functional strength training — Participants allocated to the experimental group completed three times a week, 12-week progressive resistance training protocol. This protocol consisted of functional squat system with virtual reality in leg press, plyometric exercises, exercises with Bosu ball & heel-rise exercises. This intensity of training is approximately equal to training at an intensity of 60% to 80% of one-repetition maximum according to "National Strength and Conditioning Association (NSCA)" protocols. Intensity of exercise is gradually increased 10% bi-weekly.
  Arms: intervention group

SUMMARY:
This study is aimed to investigate effectiveness of progressive functional strength training protocol (functional squat system with virtual reality in leg press, plyometric exercises, exercises with Bosu ball & heel-rise exercises) on Body Functions and activity in children with unilateral spastic Cerebral Palsy (CP) by applying current guidelines. According to literature, there are studies that investigate the effects of functional strength training in children with CP. But there is no randomized controlled trial, explore the effects of progressive functional strength training protocol on body functions and activity on unilateral spastic CP. Hypothesis of this study is that progressive functional strength training protocol improves performance-related physical fitness, gross motor function, dynamic, balance, muscle tone and muscle strength in unilateral spastic CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) describes a group of disorders in the development of movement and posture, causing activity limitations, which are attributed to non-progressive disturbances that occurred in the developing brain. It is the most common cause of movement disability in childhood. Children with CP may experience a variety of impaired muscle functions, such as spasticity, muscle weakness, and loss of selective motor control. Muscle structural changes are caused to activate of mechanisms that are limited function with growing and maturation. The weakness found in children with CP is attributable to both altered neural mechanisms and muscle tissue changes. Several factors affect the level of weakness found in the muscles of children with CP. First, weakness may differ between proximal and distal limb muscles. Stackhouse et al. found that the maximum voluntary contraction (MVC) was more impaired in the plantar flexors than the quadriceps of children with mild CP compared with controls. Second, the peak torque may vary according to the velocity of limb movement. Peak torque of the knee flexors and extensors in 24 children with CP was found to decrease with increasing velocity on an isokinetic machine. Third, peak torque may vary according to muscle length. An isokinetic study of 44 children and young people with CP found that peak torque in the hip abductors occurred when the muscle was in a lengthened position with the leg still in adduction. Fourth, the type of contraction was found to consistently affect the peak torque in both children with CP and those who are typically developing, with eccentric force being greater than concentric force in the same muscle. Although all impaired muscle functions limit the performance of daily life activities and participation in a child with CP, a recent study has shown that muscle weakness showed a stronger association with mobility limitations in children with CP than spasticity. Strength training for these children is, therefore, expected to improve or maintain their strength and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* age between 7 years and 16 years;
* classified in levels I of the Gross Motor Function Classification System (GMFCS)
* able to follow and accept verbal instructions

Exclusion Criteria:

* any orthopaedic surgery or botulinum toxin injection in the past 6 months,
* children whose parents refused to participate

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
muscle strength | change from basaline muscle strenght of lower extremities at 12 weeks
  8 channels Biopac® surface electromyography data acquisition and analysis systems for root mean square of maximum voluntary contraction, hand-held dynamometer "Power track II commander" for isometric muscle strength and functional squat rehabilitation system with leg press for one-maximum repetition was used to evaluate muscle strength.

SECONDARY OUTCOMES:
gross motor function | change from basaline gross motor funciton at 12 weeks
  Gross motor function will be assessed using dimensions D and E of the Gross Motor Function Measurement (GMFM), which consists of standing, and walking, running, and jumping. 10-metre walking and 1-minute walking will be evaluated function.
muscle tone | change from basaline muscle tone at 12 weeks
  modified Tardieu scale was used to evaluate muscle tone.
balance | change from basaline balance at 12 week
  Dynamic balance was assessed with Time up & go and functional reaching test.
functional muscle strength | change from basaline funcitonal muscle strenght at 12 weeks
  The 30s Repetition Maximum test was used to assess functional muscle strength of the lower extremities. The three closed kinetic chain exercises of lateral step-up test, sit to stand, and attain stand through half knee were used.
muscle performance | change from basaline muscle performance at 12 weeks
  Standing Broad Jump and vertical jump was used to evaluate muscle performance.
power | change from basaline short-term muscle power at 12 weeks
  Short-term muscle power was evaluated using the mean power and peak power obtained from the Muscle Power Sprint Test.
Agility | change from basaline agility at 12 weeks
  Agility was measured via using the 10x5m sprint test.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park EY, Kim WH. Meta-analysis of the effect of strengthening interventions in individuals with cerebral palsy. Res Dev Disabil. 2014 Feb;35(2):239-49. doi: 10.1016/j.ridd.2013.10.021. Epub 2013 Nov 27. PMID 24291625
- [Background] Taylor NF, Dodd KJ, Baker RJ, Willoughby K, Thomason P, Graham HK. Progressive resistance training and mobility-related function in young people with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2013 Sep;55(9):806-12. doi: 10.1111/dmcn.12190. Epub 2013 Jun 22. PMID 23789741
- [Background] Scholtes VA, Becher JG, Comuth A, Dekkers H, Van Dijk L, Dallmeijer AJ. Effectiveness of functional progressive resistance exercise strength training on muscle strength and mobility in children with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2010 Jun;52(6):e107-13. doi: 10.1111/j.1469-8749.2009.03604.x. Epub 2010 Feb 12. PMID 20132136
- [Background] Kaya Kara O, Atasavun Uysal S, Turker D, Karayazgan S, Gunel MK, Baltaci G. The effects of Kinesio Taping on body functions and activity in unilateral spastic cerebral palsy: a single-blind randomized controlled trial. Dev Med Child Neurol. 2015 Jan;57(1):81-8. doi: 10.1111/dmcn.12583. Epub 2014 Sep 12. PMID 25213082
- See also: National Strength and Conditioning Association — http://www.nsca.com/